CLINICAL TRIAL: NCT03735589
Title: A Phase I/IIa Safety and Immunologic Efficacy Trial of Intraperitoneal Induction of CTLs Combined With Alpha-Dendritic Cell Vaccine for Primary Ovarian Cancer
Brief Title: Specialized Immune Cells (nCTLs) and a Vaccine (Alpha-type-1 Polarized Dendritic Cells) in Treating Patients With Stage II-IV Ovarian, Fallopian Tube, or Primary Peritoneal Cancer
Status: Withdrawn | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: new study to be created
Sponsor: Roswell Park Cancer Institute (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: i 60417; NCI-2018-02337 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); i 60417 (Other: Roswell Park Cancer Institute); P50CA159981 (NIH)
Record Dates: First submitted 2018-11-07; First posted 2018-11-08 (Actual); Last update posted 2023-11-22 (Actual); Status verified 2023-11

CONDITIONS: Stage II Fallopian Tube Cancer AJCC v8; Stage II Ovarian Cancer AJCC v8; Stage II Primary Peritoneal Cancer AJCC v8; Stage IIA Fallopian Tube Cancer AJCC v8; Stage IIA Ovarian Cancer AJCC v8; Stage IIA Primary Peritoneal Cancer AJCC v8; Stage IIB Fallopian Tube Cancer AJCC v8; Stage IIB Ovarian Cancer AJCC v8; Stage IIB Primary Peritoneal Cancer AJCC v8; Stage III Fallopian Tube Cancer AJCC v8; Stage III Ovarian Cancer AJCC v8; Stage III Primary Peritoneal Cancer AJCC v8; Stage IIIA Fallopian Tube Cancer AJCC v8; Stage IIIA Ovarian Cancer AJCC v8; Stage IIIA Primary Peritoneal Cancer AJCC v8; Stage IIIA1 Fallopian Tube Cancer AJCC v8; Stage IIIA1 Ovarian Cancer AJCC v8; Stage IIIA2 Fallopian Tube Cancer AJCC v8; Stage IIIA2 Ovarian Cancer AJCC v8; Stage IIIB Fallopian Tube Cancer AJCC v8; Stage IIIB Ovarian Cancer AJCC v8; Stage IIIB Primary Peritoneal Cancer AJCC v8; Stage IIIC Fallopian Tube Cancer AJCC v8; Stage IIIC Ovarian Cancer AJCC v8; Stage IIIC Primary Peritoneal Cancer AJCC v8; Stage IV Fallopian Tube Cancer AJCC v8; Stage IV Ovarian Cancer AJCC v8; Stage IV Primary Peritoneal Cancer AJCC v8; Stage IVA Fallopian Tube Cancer AJCC v8; Stage IVA Ovarian Cancer AJCC v8; Stage IVA Primary Peritoneal Cancer AJCC v8; Stage IVB Fallopian Tube Cancer AJCC v8; Stage IVB Ovarian Cancer AJCC v8; Stage IVB Primary Peritoneal Cancer AJCC v8
MeSH Terms: conditions — Fallopian Tube Neoplasms; Ovarian Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- Treatment (nCTLs, alpha-DC1 vaccine) (Experimental): Patients receive the alpha-type-1 polarized dendritic cell vaccine ID 2 weeks before day 0, on day 0, and on day 28. Patients also receive aDC1 IP over 3-10 seconds on day 0. In the absence of unacceptable side effects, patients may receive the alpha-type-1 polarized dendritic cell vaccine every 1-3 months at the discretion of the physician.
  Interventions: Biological: Alpha-type-1 Polarized Dendritic Cells; Biological: Autologous Natural Killer Cell-like CTLs

INTERVENTIONS:
Biological: Alpha-type-1 Polarized Dendritic Cells — Given ID
  Other Names: alphaDC1
Biological: Autologous Natural Killer Cell-like CTLs — Given IP
  Other Names: Autologous aDC1-induced CTLs; Autologous CTLs Sensitized Ex-vivo with Autologous TAA-loaded alphaDC1; Autologous Natural Killer-like Cytotoxic Lymphocytes; Autologous nCTLs; Autologous NK-like CTLs; In Vitro DC-sensitized CTLs; n-vitro DC-sensitized Autologous CTLs; Therapeutic nCTLs; Tumor Neo-antigen-specific nCTLs

SUMMARY:
This phase I/IIa trial studies the side effects and best dose of a type of specialized immune cell (natural killer cell-like cytotoxic T-lymphocytes (CTLs) (nCTLs) and how well they work when given with a vaccine (alpha-type-1 polarized dendritic cells) in treating patients with stage II-IV ovarian, fallopian tube, or primary peritoneal cancer. nCTLs are immune cells that are isolated from each patient?s blood and "taught" in the laboratory how to recognize and eliminate tumor cells. These "educated" immune cells are then given back to the patient. An alpha-type-1 polarized dendritic cell vaccine is another population of "educated" immune cells that work to support the infused nCTLs. Giving nCTLS with a dendritic cell vaccine may work better in treating patients with ovarian, fallopian tube, or primary peritoneal cancer.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES I. To evaluate the safety, tolerability, and feasibility of intraperitoneal (i.p.) administration of autologous tumor loaded DC vaccines (alpha-type-1 polarized dendritic cell [alphaDC1]) combined with intradermally administered aDC1 .(Safety [Phase I aspect]) II. To measure the intraperitoneal induction and persistence of aDCI induced sensitized cytotoxic T Cells (CTLs), which express natural killer (NK) cell-like features (nCTLs) and total CTLs following intraperitoneal administration of aDC1. (Local Immunologic Efficacy [Phase II aspect])

SECONDARY OBJECTIVES I. To study the T cell populations generated that correlates with higher anti-tumor responses.

EXPLORATORY OBJECTIVES I. To evaluate the progression-free survival and overall survival of patients treated with this regimen.

OUTLINE: This is a phase I, dose-escalation study of nCTLs, followed by a phase IIa study.

Patients receive the alpha-type-1 polarized dendritic cell vaccine intradermally (ID) 2 weeks before day 0, on day 0, and on day 28. Patients also receive nCTLs intraperitoneally (IP) over 15-30 minutes on day 0. In the absence of unacceptable side effects, patients may receive the alpha-type-1 polarized dendritic cell vaccine every 1-3 months at the discretion of the physician.

After completion of study treatment, patients are followed up at 14 days, then at 6 and 12 months.

ELIGIBILITY:
Inclusion Criteria:

* Eligible patients will be women with stages II-IV epithelial ovarian, fallopian tube, or primary peritoneal carcinoma with no radiologic evidence of disease (NED) or minimal disease burden after 1st line therapy. These patients would normally enter a period of observation after standard management.
* Life expectancy > 6 months.
* Have been informed of other treatment options.
* Patients must be reasonable candidates for intraperitoneal (IP) port placement with no prior evidence of persistent abdominal wall or intraperitoneal infections, renal toxicity, or bowel obstruction or fistula.
* Patients must have documented available tumor: at least 1 cm of bulk tumor mass collected at the time of primary or interval debulking surgery. The specimen may be obtained on this protocol or as part of other Institutional Review Board (IRB) approved tumor banking protocols.
* Patients should be free of active infection requiring antibiotics (with the exception of uncomplicated urinary tract infection [UTI]).
* Must have adequate venous access for apheresis. (Pheresis catheter placement for cell collection is allowed).
* Patient must agree to leukapheresis.
* Patients must agree to appropriate clinical monitoring to receive the study regimens.
* Absolute neutrophil count (ANC) greater than or equal to 1,000/uL.
* Platelets greater than or equal to 75,000/uL.
* Hemoglobin greater than or equal to 8.0 g/dL.
* Creatinine less than or equal to 2 x institutional upper limit normal (ULN).
* Bilirubin less than or equal to 1.5 x ULN.
* Serum glutamic oxaloacetic transaminase (SGOT) less than or equal to 3 x ULN.
* Alkaline phosphatase less than or equal to 3 x ULN.
* Participant or legal representative must understand the investigational nature of this study and sign an Independent Ethics Committee/Institutional Review Board approved written informed consent form prior to receiving any study related procedure.
* Female subjects must either be of non-reproductive potential (i.e., post-menopausal by history: >= 50 years old and no menses for >= 1 year without an alternative medical cause; OR history of hysterectomy, OR history of bilateral tubal ligation, OR history of bilateral oophorectomy) or must have a negative urine or serum pregnancy test within 28 days of study treatment, confirmed prior to treatment.
* Patients must have an Eastern Cooperative Oncology Group (ECOG) Performance Status of 0 or 1.

Exclusion Criteria:

* Metastatic disease to the central nervous system and any site above diaphragm.
* Other serious illnesses (e.g., serious infections requiring antibiotics [with the exception of uncomplicated UTI], bleeding disorders).
* Chemotherapy, radiation therapy, or immunotherapy within 4 weeks prior to first dosing of study agent. Concomitant hormonal therapies are allowed.
* Patients who have an active autoimmune disease (e.g., rheumatoid arthritis, systemic lupus erythematosus [SLE], ulcerative colitis, Crohn's Disease, multiple sclerosis [MS], ankylosing spondylitis) requiring chronic use of steroids or other immunosuppressives.
* Patients being chronically treated with immunosuppressive drugs such as cyclosporin, adrenocorticotropic hormone (ACTH), or systemic chronic corticosteroids. NOTE: Recent or current use of inhaled steroids is not exclusionary.
* Use of chronic corticosteroids, hydroxyurea, or immunomodulating agents (e.g., interleukin 2, interferon alpha or gamma, granulocyte colony stimulating factors, etc.) within 30 days prior to study entry.

  * NOTE: Recent or current use of inhaled steroids is not exclusionary. If subjects are prescribed a brief course of oral steroids, the use should be limited to less than 7 days. Use of steroids before apheresis and immune assessment blood draws will affect white blood cell function (wash out period of 1 week).
* Patients with a known immunodeficiency disease including cellular immunodeficiencies, hypogammaglobulinemia or dysgammaglobulinemia; patients who have acquired, hereditary, or congenital immunodeficiencies. Specific testing is not required, however may be done as clinically indicated.
* Patients with uncontrolled diseases other than cancer may be excluded if after consultation with PI and research team it is decided it might affect the treatment efficacy or toxicity..
* Patients with tumors of low malignant potential, except ovarian pseudomyxoma or with no peritoneal disease at initial diagnosis.
* Patients with a history of other invasive malignancies, with the exception of nonmelanoma skin cancer, are excluded if there is any evidence of other malignancy being present within the last three years. Patients are also excluded if their previous cancer treatment contraindicates this protocol therapy.
* Evidence of current drug or alcohol abuse or psychiatric impairment, which in the investigator's opinion will prevent completion of the protocol therapy or follow-up. Specific testing is not required, however may be done as clinically indicated.
* Any condition that in the opinion of principal investigator (PI) would preclude patient from successfully completing the protocol therapy or follow-up.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2023-12-15 (Estimated); Primary Completion 2025-12-01 (Estimated); Study Completion 2025-12-01 (Estimated)

PRIMARY OUTCOMES:
Incidence of adverse events as assessed by Cancer Therapy Evaluation Program (CTEP) version 4 of the Common Terminology Criteria for Adverse Events (CTCAE) | Up to 12 months
Dose-limiting toxicities (DLT) assessed by CTCAE version 5 | Up to 14 days after intraperitoneal (IP) infusion of nCTLs
  Will be used in the estimation of the maximum tolerated dose (MTD) and the accompanying of the dose escalation decisions. However, no formal analyses of DLTs are planned.
Change in immune response | From baseline (day 0) to day 2 (48 hours after adoptive cell therapy [ACT]) administration
  Change in immune response will be measured by the increase in the number of CD3+CD8+NKG2D (high) natural killer cell-like cytotoxic T-lymphocyte (CTLs) (nCTLs) and the increase in total CD3+CD8+ CTLs recovered in the peritoneal washes with evaluation on day 0 versus day 2. The analysis will consist of an analysis-of-covariance (ANCOVA) for the outcome of post-pre ACT treatment cell count with a factor for dose and sampling time 48 hrs +/- 24 hrs.
Persistence of nCTLs after their adoptive transfer | Up to 4 weeks
  At day 0 will obtain peritoneal material (outflow and washes) directly before i.p. infusion of nCTLs, as well as day 2 (48 hours +/- 24 hours), day 7 (+/- 2 days), 2 weeks (14 days +/- 2 days) and 4 weeks (28 days +/- 3 days) later.

SECONDARY OUTCOMES:
T cell populations and higher anti-tumor responses | Up to 4 weeks
  Will estimate the half-life of CD3/CD8/NKG2D (triple-positive nCTLs) cell counts and longitudinal changes CD3/CD8 cell counts (double-positive CTLs, which include both nCTLs and additional CTLs newly recruited CTLs from the circulation) cell counts as a function of dose and time. A nonlinear regression model with a random effect for subject (population pharmacokinetics [PK]) will be fit to a one-compartment kinetics first-order absorption model per dose level.

OTHER OUTCOMES:
Progression-free survival assessed by immune-related response criteria (irRECIST) | Up to 12 months
  Will examine time-to-disease progression graphically via the generation of Kaplan-Meier survival curves.
Overall survival assessed by irRECIST | Up to 12 months
  Will examine time-to-disease progression graphically via the generation of Kaplan-Meier survival curves.

CONTACTS AND LOCATIONS:
Overall Officials: Emese Zsiros, MD, PhD, Principal Investigator — Roswell Park Cancer Institute
Locations (1):
- Roswell Park Cancer Institute, Buffalo, New York, United States